CLINICAL TRIAL: NCT04144790
Title: Impact of Iron Supplementation Treatment on Brain Iron Concentrations Among Children With ADHD & Restless Leg Syndrome Combined With Periodic Limb Movements in Sleep
Brief Title: Impact of Iron Supplementation Treatment on Brain Iron Concentrations
Status: Completed | Type: Observational
Sponsor: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: KKI
Record Dates: First submitted 2019-10-27; First posted 2019-10-30 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: ADHD; Iron-deficiency; Restless Legs Syndrome; Periodic Limb Movement Sleep Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Anemia, Iron-Deficiency; Restless Legs Syndrome | interventions — ferrous sulfate

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ADHD+RLS: Twelve participants between the ages of 5 and 18 years with a clinical diagnosis of either RLS or ADHD, and iron deficiency.
  Interventions: Dietary Supplement: ferrous sulfate

INTERVENTIONS:
Dietary Supplement: ferrous sulfate — Although established guidelines do not currently exist for iron supplementation for children, studies have demonstrated effectiveness of a 3-month treatment regimen of 5mg/kg per day of orally-administered ferrous sulfate in reducing PLMS and subjective RLS symptoms and in increasing serum ferritin levels. Ferrous sulfate 80 mg/day resulted in improvement of ADHD symptoms in iron-deficient children.

SUMMARY:
The goal of the present study is to provide novel data to evaluate brain iron concentration as a mediator of the association between iron supplementation treatment and improvement in symptoms of ADHD and RLS in children, including PLMS. Twelve participants between the ages of 10 and 15 years will be recruited via Kennedy Krieger Institute's Sleep Disorders Clinic. Eligible participants will be asked to complete, at baseline (pre-iron supplementation treatment) and again at follow-up (post-treatment): 1) a 7 Tesla MRI scan, 2) five consecutive nights of RestEaZe™ monitoring, 3) caregiver-reported (or patient-reported if over the age of 10 years) International Restless Leg Syndrome Scale (IRLSS), and 4) caregiver-reported ADHD Rating Scale-5. The treatment interval will be 3 months.

DETAILED DESCRIPTION:
The goal of the present study is to provide novel data to evaluate brain iron concentration as a mediator of the association between iron supplementation treatment and improvement in symptoms of ADHD and RLS in children, including PLMS. Aim 1 is to evaluate the impact of iron supplementation treatment on peripheral iron concentrations and brain iron concentrations. The investigators hypothesize that iron supplementation treatment will result in increased peripheral and brain iron concentrations. Aim 2 is to evaluate the impact of iron supplementation treatment on symptoms of ADHD and restlessness during sleep. The investigators hypothesize that iron supplementation treatment will result in decreased symptoms of ADHD and restlessness during sleep. Aim 3 is to investigate the relation between brain iron concentrations and symptoms of ADHD and restlessness during sleep, including PLMS. The investigators hypothesize that brain iron concentrations in the substantia nigra and in the thalamus will be negatively related to symptoms at baseline. Aim 4 is to evaluate whether brain iron concentrations mediate the association between iron supplementation treatment and symptoms of ADHD and restlessness during sleep. The investigators hypothesize that increases in brain iron concentrations in the substantia nigra and in the thalamus will fully explain any improvements in symptoms that occur with iron supplementation treatment.

Twelve participants between the ages of 10 and 15 years will be recruited via Kennedy Krieger Institute's Sleep Disorders Clinic. Recruitment will be accomplished by posting flyers with study information at the clinic and by asking Sleep Disorders Clinic clinicians to discuss the study with their patients who may be eligible and their caregivers. In order to be included in the study, participants will need to have: 1) a clinical diagnosis of ADHD, 2) parent or patient self report of restless sleep, 3) serum iron values with ferritin < 50 mcg/L . Exclusionary criteria will be: 1) family is not proficient in English language, 2) child is in foster care, 3) child has a chronic medical condition or genetic/metabolic disorder that might impact iron metabolism, 4) child has another sleep disorder or neuropsychiatric condition that might influence sleep, RLS, or ADHD symptoms, and 6) child has been receiving iron supplementation or a medication that could disrupt sleep.

An uncontrolled open label trial design is proposed for this pilot study, in order to establish evidence to support a larger blinded, placebo-controlled trial application. Eligible participants will be asked to complete, at baseline (pre-iron supplementation treatment) and again at follow-up (post-treatment): 1) a 7 Tesla MRI scan, 2) five consecutive nights of RestEaZe™ monitoring, 3) caregiver-reported or patient-reported if over the age of 10 years International Restless Leg Syndrome Scale (IRLSS), and 4) caregiver-reported ADHD Rating Scale-5. The treatment interval will be 3 months, which has been sufficient in previous studies to allow for treatment effects to be observed. Investigators anticipate 20 to 30% attrition over the course of the 3 months of treatment, leaving 8-10 participants to scan at follow-up.

ELIGIBILITY:
Inclusion Criteria:

* a clinical diagnosis of RLS
* a clinical diagnosis of ADHD
* PLMS > 3/hour, based on average of 5 nights of home recording with RestEaze leg meters
* fasting serum iron values with ferritin < 50 mcg/kg and transferrin saturation < 45%

Exclusion Criteria:

* family is not proficient in English language
* child is in foster care
* child has a chronic medical condition or genetic/metabolic disorder that might impact iron metabolism
* child has another sleep disorder or neuropsychiatric condition that might influence sleep, RLS, or ADHD symptoms
* child has been receiving iron supplementation, psychostimulant treatment, or a dopamine agonist within the past 6 months.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Twelve participants between the ages of 5 and 18 years will be recruited via Kennedy Krieger Institute's Sleep Disorders Clinic. Recruitment will be accomplished by posting flyers with study information at the clinic and by asking Sleep Disorders Clinic clinicians to discuss the study with their patients who may be eligible and their caregivers.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Change in ADHD symptoms | Change from pre- to post- 3 months of iron supplementation treatment
  Change in ADHD symptoms measured by parent-reported ADHD-RS-V
Change in RLS symptoms | Change from pre- to post- 3 months of iron supplementation treatment
  Change in RLS symptoms measured by and RestEaZe™ monitors

SECONDARY OUTCOMES:
Change in brain-based iron concentrations | Change from pre- to post- 3 months of iron supplementation treatment
  Change in brain-based iron concentrations indexed by 7 Tesla MRI scans
Change in blood-based iron concentrations | Change from pre- to post- 3 months of iron supplementation treatment
  Change in blood-based iron concentrations indexed by ferritin and transferrin

CONTACTS AND LOCATIONS:
Overall Officials: Alison E Pritchard, PhD, Principal Investigator — Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Locations (1):
- Kennedy Krieger Institute, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
Unknown at this time